CLINICAL TRIAL: NCT06741735
Title: Study of Fetal Health Outcomes: Working With a Missouri E-telehealth Platform
Brief Title: Study of Fetal Health Outcomes: Working With a Missouri E-telehealth Platform (The SHOW-ME Study)
Acronym: SHOW-ME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Missouri, Kansas City (Other); Affinia Healthcare (Unknown)
Responsible Party: Principal Investigator, Karen Florio, Obstetrician/Gynecologist (DO MPH), University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2097887
Record Dates: First submitted 2024-12-10; First posted 2024-12-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: Non-stress test; Home Fetal Monitoring; Telehealth; High-risk Pregnancy; Social determinants of health; Cost-effectiveness; NUVO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- At-home fetal monitoring (Experimental): Participants in this arm will be prescribed an INVU at-home fetal monitoring system. All training on the device use, troubleshooting, and accessing the cloud platform for telehealth (fetal) visits will be done by INVU through the INVU app. Non-stress testing will be done from home once or twice weekly as determined by provider at scheduled date and times.
  Interventions: Device: INVU fetal monitoring system
- In-office fetal monitoring (No Intervention): In this arm, typical standard of care in-office fetal monitoring visits will be done. Participants will have non-stress testing done in clinic once or twice weekly as determined by provider at scheduled date and times.

INTERVENTIONS:
Device: INVU fetal monitoring system — INVU fetal monitoring system allows for at-home non-stress testing as opposed to the typical in-clinic testing
  Arms: At-home fetal monitoring

SUMMARY:
The goal of this clinical trial is to evaluate the potential benefit to patients and providers from using the remote fetal-monitoring system NUVO along with its app to allow for pregnant patients requiring weekly non-stress testing to do so from their homes. The main questions the investigators are looking to answer are:

What effect does the NUVO remote fetal monitoring system have on patient/provider satisfaction?

What is the cost savings (both direct and indirect) from using a remote fetal monitoring system as opposed to in-person testing for both the patient and the provider?

Researchers will compare the survey responses by both patients and providers for pre and post implementation of the NUVO fetal monitoring system to the survey responses of patients and providers who used the traditional in-clinic method to evaluate satisfaction and cost savings.

Participants will:

Answer pre-implementation surveys before undergoing the trial

Be randomly assigned to do either fetal testing at-home or in-clinic once or twice weekly as up to the provider

Before hospital discharge or within the last office visit participants will be given a post-implementation survey

DETAILED DESCRIPTION:
The goal of the investigators is to study aspects of the implementation of a new, FDA-approved technology and conduct quantitative analyses to describe reach and patient-centered predictors of use (e.g. transportation barriers), as well as qualitative analyses (i.e. focus groups with patients and providers). Focus groups were previously performed with participants randomly recruited at each institution to inform the pre-implementation questionnaires for the patients.

For this study, participants will be identified through their PIs institution, as someone who is 18 years of age or older, who has been identified by their providers as someone who requires antenatal fetal testing (starting at 32 weeks), and who has a smart device with WIFI access. Participants with Medicaid insurance will have their expenses covered by insurance as currently Medicaid covers the cost of home fetal telehealth. Participants who are self-pay or who have private insurance will be offered to participate but informed that they will have to pay all expenses out of pocket (as currently in Missouri private payers are not reimbursing for the use of home fetal monitors). All participants will be required to sign an informed consent prior to enrollment.

Questionnaires were iteratively designed by the PIs at each institution. Pre-implementation questionnaires will be distributed to eligible patients and provider (including nurses, Medical Assistants, and scheduling Staff)) enrolled at all 3 centers. Patient participants will be approached between 12-28 weeks and must meet the inclusion criteria outlined below. Providers will be approached prior to the start of enrollment at each institution to discuss their desire to read INVU NSTs remotely as part of the study and will be consented at that time. Providers are eligible if they are board certified or eligible in family medicine, obstetrics and gynecology, or maternal-fetal medicine and read NSTs as part of their routine care delivery to obstetrical patients. Nurse practitioners who provide obstetrical care and are qualified to read NST (as part of routine care), Nurses, Medical Assistants, and Scheduling staff are also eligible to participate as a provider. Eligibility will be verified prior to enrollment. Patient eligibility will be verified prior to enrollment. Following, subjects will be asked whether or not they want to participate in the fetal testing portion of the study. For those who desire to perform the in-home fetal monitoring, they will then be randomized in a 1:1 manner to either in office or home monitoring. Although not testing the effectiveness of the device itself, randomization will ensure that investigators prevent inclusion bias (inherit differences that may be present between those who do not choose to participate and those who do participate) by having all those who want to participate randomly assigned to either receive in-home testing or in-office testing. For those in the home monitoring group, a prescription for the device will be given and the equipment will be shipped to the participants home within 6-10 business days. All training on the device use, troubleshooting, and accessing the cloud platform for telehealth (fetal) visits will be done by INVU through the INVU app. INVU provides an effective, easy-to-use chat service within the application for customer support for these training sessions. A number as well as printed instructions for troubleshooting will be provided to each enrolled individual for easy, 24-hour access to INVU at home. For participants who are randomized to the in-office monitoring, they will continue their standard of care monitoring as they would regardless of being part of the study. The testing and frequency itself will not differ between the groups (i.e. all participants will still receive non-stress testing once or twice weekly as determined by their provider) rather just the location (i.e. in home or in office). Participants will be scheduled as they would normally and will have specified times to place the band and start their fetal monitoring session. Since INVU is not part of routine clinical care at any of the current institutions, participants who choose not to be part of the study will not have the opportunity to use INVU outside of the study.

The routine clinical care group will maintain their obstetrical care as prescribed by their provider and will continue their antenatal fetal testing in the office or hospital setting. They will not be asked to provide any additional testing or information (i.e. questionnaires) after randomization. Investigators will be collecting demographic and clinical outcomes information, including costs at the end of study.

For the at-home fetal monitoring portion, this study will be utilizing "INVU" technology designed by Nuvo to perform fetal testing remotely. As the patient will not be in the ambulatory setting and part of routine antenatal testing includes maternal vital signs, investigators will be providing the at-home participants with blood pressure cuffs (through prescription, or as part of the free Cuff Kit project if available at participating institutions) so they can monitor their blood pressure.

"INVU™ is the first FDA-cleared remote pregnancy monitoring platform that allows expectant mothers to monitor maternal and fetal health from anywhere under the supervision of their physician. INVU is a maternal-fetal monitor that non-invasively measures and displays fetal heart rate (FHR) and maternal heart rate (MHR). The INVU acquires and displays the FHR and MHR tracings from abdominal surface electrodes that pick up the fetal and maternal heart biopotential signals as well as acoustic phonocardiogram signals. Unlike current FHR monitoring, INVU does not utilize Doppler or traditional tocometer technology, and is therefore not dependent on monitor placement, maternal body habitus, fetal movement and presentation, or maternal positioning. The INVU system is composed of a wearable sensor band with multiple sensors, coupled to a mobile device with the appropriate applications for control and display of the results, and a bridge that connects to cloud-based applications, which perform signal processing, patient/doctor database management and data storage. In addition to the INVU monitor, INVU is paired with a mobile application available to iOS and Android users. The INVU application provides the pregnant individual real-time information regarding the fetal heart rate and can only be used during the previously agreed-upon visit time. Maternal data collected will include blood pressure, that is collected via an approved cuff provided (either through their insurance company or through the Cuff Kit project) and distributed at the time of enrollment. These blood pressures will automatically upload into the INVU app through blue-tooth technology. The patients will be asked to take their blood pressure at home during their NST visit according to standard of care. For instance, if it is the standard of care at one institution to monitor blood pressure with each NST, this will be done in the patient's home and reported at the time of her telehealth visit with the doctor. It will either be verbally reported or, in the event there is no telehealth visit scheduled with the NST, it will be uploaded to the INVU platform for review by the provider when the NST is read. Any abnormal readings will be handled according to the standard of care at each institution. The data will be collected and communicated to an approved provider. Frequency and type of monitoring (i.e. fetal non-stress test versus biophysical profile) will be according to institutional protocols and provider preference; this study will not determine level of care required.

According to each institution's standard of care, the participant will be assigned a "visit" time when she/he/they will be instructed to place the device and turn on the smart device. Prior to enrollment, questions on access to smart devices and WIFI will be asked in order to assess reliability of adhering to the testing regimen. In the event a patient's Wi-Fi is not functional, he/she/they will be asked to come to an in-person appointment at the office instead to complete her exam, on a date that is mutually agreed upon between the provider and the patient. At the designated time, the patient will perform the NST and according to workflow within each institution, the output will be interpreted. At the end of the pregnancy, all the equipment will be sent back to the company in a pre-package, stamped box. Once the device is received, the participants in the INVU group will receive a $50 gift card by email or at their next clinic appointment (if any remain following antenatal testing), whichever is most convenient for them. Prior to discharge from the hospital or at last in-office visit, participants will be provided a post-implementation questionnaire. Those who were part of the control group (ambulatory monitoring or standard of care) will receive their gift card at confirmation of delivery and discharge from the hospital. Providers will not be eligible for a gift card as part of this study.

All clinical data will be integrated and uploaded into the electronic medical record. NST readouts can be scanned directly into the EMR in PDF form. All research-appropriate data will be entered and stored in a password-protected, hospital network database (REDcap) in the primary PIs office.

ELIGIBILITY:
Inclusion Criteria

* English Speaking
* > 18 years of age
* Singleton gestation
* Missouri Medicaid as primary insurance (paid by study), offered to patients with private insurance for self-pay
* Requires antenatal testing between 32-40 weeks according to institutional policies
* One of the following indications for fetal NST:

  * Gestational diabetes
  * Well-controlled type II diabetes
  * Chronic hypertension without evidence of placental insufficiency
  * Advanced maternal age
  * Obesity (as defined as BMI >30 and <45)
* Android or iOS system-operated telephone or tablet
* Home or work access to reliable internet (WIFI screening completed by research personnel)

Exclusion Criteria

* Multiple gestations
* Additional co-morbidities not listed in the inclusion criteria
* PPROM or evidence of preterm labor
* Oligohydramnios of < 5 cm of polyhydramnios > 30
* Co-existing fetal complications: FGR, placenta or vasa previa, fetal chromosomal or structural anomaly, recent (within a week) fetal testing of a BPP < 8/10 prior to enrollment
* Intention to transfer care to different provider during the pregnancy
* Currently institutionalized or incarcerated
* Inability to consent for oneself
* <18 years of age
* History of prior stillbirth
* Lack of access to reliable internet
* Abdominal skin disorder that prevents use of the INVO device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the implementation of a remote fetal-monitoring system through RE-AIM quest framework | Participants will be recruited at any time during pregnancy if they meet inclusion criteria and require antenatal fetal testing between 32 and 40 weeks gestation
  Each of the three participating centers and patients will receive access to and training in the INVU telehealth platform with the goal of studying the implementation (through pre and post implementation questionnaires) of this novel telehealth system and its impact on both patients and providers

SECONDARY OUTCOMES:
Assess direct and indirect cost savings for patients, providers, and insurance carriers following implementation of a remote monitoring system | Participants will be recruited at any time during pregnancy if they meet inclusion criteria and require antenatal fetal testing between 32 and 40 weeks gestation
  Investigators will evaluate cost savings by numerating averted emergency room, triage, facility fees, and office visits for fetal symptoms (i.e. decreased fetal movement). Furthermore, investigators will assess cost savings for patients by numerating facility fees, transportation costs, and utilization of hospital resources for those utilizing the home monitoring system as compared to participants who received ambulatory evaluation.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Missouri, Columbia, Missouri
  - University of Missouri - Kansas City, Kansas City, Missouri
  - Affinia Healthcare, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified. No participant data will be shared

REFERENCES:
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Arias MP, Wang E, Leitner K, Sannah T, Keegan M, Delferro J, Iluore C, Arimoro F, Streaty T, Hamm RF. The impact on postpartum care by telehealth: a retrospective cohort study. Am J Obstet Gynecol MFM. 2022 May;4(3):100611. doi: 10.1016/j.ajogmf.2022.100611. Epub 2022 Mar 22. PMID 35331971
- [Background] Muppavarapu K, Saeed SA, Jones K, Hurd O, Haley V. Study of Impact of Telehealth Use on Clinic "No Show" Rates at an Academic Practice. Psychiatr Q. 2022 Jun;93(2):689-699. doi: 10.1007/s11126-022-09983-6. Epub 2022 Apr 12. PMID 35412100
- [Background] Hoppe KK, Thomas N, Zernick M, Zella JB, Havighurst T, Kim K, Williams M, Niu B, Lohr A, Johnson HM. Telehealth with remote blood pressure monitoring compared with standard care for postpartum hypertension. Am J Obstet Gynecol. 2020 Oct;223(4):585-588. doi: 10.1016/j.ajog.2020.05.027. Epub 2020 May 19. No abstract available. PMID 32439388
- [Background] Aziz A, Zork N, Aubey JJ, Baptiste CD, D'Alton ME, Emeruwa UN, Fuchs KM, Goffman D, Gyamfi-Bannerman C, Haythe JH, LaSala AP, Madden N, Miller EC, Miller RS, Monk C, Moroz L, Ona S, Ring LE, Sheen JJ, Spiegel ES, Simpson LL, Yates HS, Friedman AM. Telehealth for High-Risk Pregnancies in the Setting of the COVID-19 Pandemic. Am J Perinatol. 2020 Jun;37(8):800-808. doi: 10.1055/s-0040-1712121. Epub 2020 May 12. PMID 32396948